CLINICAL TRIAL: NCT03124433
Title: Neoadjuvant Apalutamide (ARN509) and Radical Prostatectomy in the Treatment of Intermediate to High Risk Prostate Cancer
Brief Title: Neoadjuvant Apalutamide (ARN509) and Radical Prostatectomy in Treatment of Intermediate to High Risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARN509 - 2016
Record Dates: First submitted 2017-04-09; First posted 2017-04-21 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Cancer of the Prostate
Keywords: prostate cancer; prostatectomy, retropubic; Androgen Receptor Antagonists
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant apalutamide (Experimental): Oral apaluatmide 240mg daily for 12 weeks followed by standard of care robotic radical prostatectomy and pelvic node dissection
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Participants will receive oral apalutamide 240mg daily for 12 weeks
  Other Names: ARN509

SUMMARY:
This is an investigator-initiated phase II single arm trial, combining neoadjuvant apalutamide (ARN509) with radical prostatectomy, in the treatment of D'Amico intermediate to high risk organ-confined prostate cancer. Apalutamide has shown efficacy in castrate resistant prostate cancer in phase II studies and are now in phase III trials combined with radiation in organ confined disease.

The primary study objectives include assessment of (i) oncological efficacy as determined by tumour downstaging and achievement of nadir PSA The secondary study objectives include(i) determination of adverse effects related to apalutamide and surgical complication rates (ii) human prostate tissue effect of apalutamide

The study will recruit thirty eligible participants who will receive 12 weeks of oral apalutamide 240mg daily. This will be followed by standard-of-care radical prostatectomy. The total trial duration is 26 weeks.

DETAILED DESCRIPTION:
This is a phase II single arm study looking at the efficacy of 12 weeks of neoadjuvant apalutamide (ARN 509), combined with standard-of-care radical prostatectomy, for D'Amico intermediate to high risk prostate cancer patients. The phases of the study will include: screening, treatment and follow-up phases.

Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed primary adenocarcinoma of the prostate gland
* non-metastatic D'Amico intermediate to high risk patients undergoing radical prostatectomy as primary definitive therapy
* no known hypersensitivity to the study drug
* able to swallow study drug as whole tablets

Exclusion Criteria:

* presence of small cell, neuroendocrine or ductal differentiation at needle biopsy
* individuals with prior pelvic irradiation therapy for any form of pelvic malignancy
* patients with psychiatric conditions requiring anti-psychotic therapy, or preventing the provision of informed consent
* renal impairment with serum creatinine more than twice the upper limit of normal
* Other prior malignancy less than or equal to 5 years prior to recruitment
* ECOG performance status 2 or poorer

Ages: 21 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with pathological downstaging after neodjuvant apalutamide followed by radical prostatectomy | 24 weeks
  This is described as residual cancer burden and treatment response group on histopathology after neoadjuvant apalutamide and radical prostatectomy
Proportion of patients with biochemical treatment response following neoadjuvant apalutamide and radical prostatectomy | 24 weeks
  Patients who attain serum PSA levels below 0.03microg/L

SECONDARY OUTCOMES:
Proportion of patients who report significant adverse effects after 12 weeks of neoadjuvant apalutamide | 12 weeks
  Adverse effects as defined by CTCAE criteria grade 3 and above
The proportion of patients with peri-operative complications following neoadjuvant apalutamide and radical prostatectomy | 24 weeks
  The level of complications defined by Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Lui Shiong Lee, MBBS,MRCS, Principal Investigator — Singapore General Hospital
Locations (1):
- Department of Urology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang X, Allen JC, Aslim EJ, Tay KJ, Yuen SPJ, Kanesvaran R, Chua MLK, Chong TW, Ho SSH, Lee LS. Patient-reported outcomes of a phase II neoadjuvant apalutamide (ARN-509) and radical prostatectomy in treatment of intermediate- to high-risk prostate cancer (NEAR) trial. Int J Urol. 2022 Nov;29(11):1322-1330. doi: 10.1111/iju.14994. Epub 2022 Aug 24. PMID 36000794
- [Derived] Lee LS, Sim AYL, Ong CW, Yang X, Ng CCY, Liu W, Rajasegaran V, Lim AMS, Aslim EJ, Ngo NT, Khor LY, Kanesvaran R, Allen JCJ, Tay KJ, Yuen JSP, Chong TW, Ho SSH, Teh BT, Chua MLK. NEAR trial: A single-arm phase II trial of neoadjuvant apalutamide monotherapy and radical prostatectomy in intermediate- and high-risk prostate cancer. Prostate Cancer Prostatic Dis. 2022 Apr;25(4):741-748. doi: 10.1038/s41391-022-00496-8. Epub 2022 Jan 28. PMID 35091711